CLINICAL TRIAL: NCT01157494
Title: Validity of Manipulation Taxonomy of Spastic Hemiplegic Cerebral Palsy Forms Proposed by Ferrari A et.al.
Brief Title: Validity of Manipulation Taxonomy of Spastic Hemiplegic Cerebral Palsy (CP) Forms
Status: Completed | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Collaborators: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Adriano Ferrari, University of Modena and Reggio Emilia and Hospital Azienda Santa Maria Nuova Reggio Emilia
Other Study IDs: UDGEE_2010_hand_class
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-04

CONDITIONS: Hemiplegia; Cerebral Palsy
Keywords: cerebral palsy; hemiplegia; upper limb; assessment; classification system
MeSH Terms: conditions — Hemiplegia; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- children with hemiplegia: To determine the criterion validity of the classification of the pattern of manipulation proposed by Ferrari et al. we correlated hand manipulation classes with both the scores of the two standard criteria chosen (AHA and Melbourne Assessment).
  Interventions: Other: classification of hand manipulation function

INTERVENTIONS:
Other: classification of hand manipulation function — To determine the criterion validity of the classification of the pattern of manipulation proposed by Ferrari et al. we correlated hand manipulation classes with both the scores of the two standard criteria chosen (AHA and Melbourne Assessment).

SUMMARY:
In recent years Ferrari et al. proposed a new classification of manipulation in children with spastic hemiplegia which describes five different classes by analyzing and integrating the kinematic patterns of the hand and its functional use.

The investigators believe that this classification provides the clinician with clinically meaningful information, by identifying the useful strategies spontaneously adopted by the children during manipulation tasks.

The aim of this study is to determine the criterion validity of the new classification of the pattern of manipulation in children with spastic hemiplegia by correlating hand manipulation classes with both the scores of the Assisting Hand Assessment and the scores of the Melbourne Assessment of Unilateral Upper Limb Function.

ELIGIBILITY:
Inclusion criteria:

* clinical and instrumental (TC or RMN) diagnosis of child hemiplegia
* age > 5 years

Exclusion criteria:

* acquired hemiplegia at the age > 3 years
* anti-spastic drug inoculations or functional surgery on the plegic UE 6 months prior to the video recordings
* severe mental retardation attested by the Diagnostic and Statistical Manual of mental disorders IV
* pharmaco-resistant epilepsy
* behavioural disorders

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We retrospectively studied children with hemiplegia and CP who are followed by the Unit for Severe Disability in the Developmental Age at the Hospital of Reggio Emilia (Italy).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Assisting Hand Assessment (AHA) | the 2 assessment has to be registered within 6 months
  correlation between the new classification of hand manipulation function and the AHA which measures the bi-manual performance, i.e. what the child usually does with the plegic hand

SECONDARY OUTCOMES:
Melbourne Assessment of Unilateral Upper Limb Function (Melbourne Assessment) | the 2 assessment has to be registered within 6 months
  correlation between the new classification of hand manipulation function and the Melbourne Assessment which measures the bi-manual performance, i.e. what the child usually does with the plegic hand

CONTACTS AND LOCATIONS:
Overall Officials: Adriano Ferrari, MD, Study Chair — University of Modena and Reggio Emilia and Hospital Santa Maria Nuova; Giulia Borelli, PT, Principal Investigator — Azienda USL Reggio Emilia
Locations (1):
- Hospital Azienda Santa Maria Nuova in Reggio Emilia, Reggio Emilia, RE, Italy